CLINICAL TRIAL: NCT00532961
Title: A Randomized, Double-masked, Parallel Comparison of Ocular Tolerance and IOP Effects of Zylet vs TobraDex Administered Four Times Daily for Four Weeks in Healthy Volunteers
Brief Title: Ocular Tolerance and Intraocular Pressure (IOP) Effects of Zylet Versus Tobradex
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 372
Record Dates: First submitted 2007-09-20; First posted 2007-09-21 (Estimated); Last update posted 2011-12-08 (Estimated); Status verified 2011-12

CONDITIONS: Inflammation
MeSH Terms: conditions — Inflammation | interventions — Loteprednol Etabonate; Dexamethasone; Tobramycin, Dexamethasone Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Zylet (Experimental): Zylet (loteprednol etabonate and tobramycin)
  Interventions: Drug: Loteprednol etabonate 0.5% and tobramycin 0.3%
- Tobradex (Active Comparator): TobraDex (dexamethasone and tobramycin)
  Interventions: Drug: Dexamethasone 0.1% and tobramycin 0.3%

INTERVENTIONS:
Drug: Loteprednol etabonate 0.5% and tobramycin 0.3% — ophthalmic suspension, four times daily during the day at roughly 4 hour intervals(1-2 drops per eye)for a total of 28 days
  Other Names: Zylet
  Arms: Zylet
Drug: Dexamethasone 0.1% and tobramycin 0.3% — ophthalmic suspension, four times daily during the day at roughly 4 hour intervals (1-2 drops/eye) for a total of 28 days.
  Other Names: TobraDex
  Arms: Tobradex

SUMMARY:
Phase IV, randomized, double-masked, parallel-group clinical trial comparing the ocular tolerability and steroid-induced intraocular pressure (IOP) effects of Zylet wth that of TobraDex in healthy volunteers, when either product was administered QID (at approximately 4-hour intervals) for 28 days.

ELIGIBILITY:
Inclusion Criteria:

* in good general health based on investigator judgment
* able and willing to follow instructions, provide informed consent, make the required study visits, and use an electronic patient diary during the study
* possessing a best corrected visual acuity of at least 20/40 in each eye
* for females, using reliable contraception and a negative urine pregnancy test prior to study entry

Exclusion Criteria:

* contact lenses worn within 30 days prior to enrollment or during study period
* known hypersensitivity to study medication or any component
* presence of significant ocular or systemic disease that might interfere with the interpretation of the results
* a need for administration of chronic topical ocular or systemic medications of any kind during the study.
* participation in an opthalmic drug or device research study within 30 days prior to entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2005-02; Primary Completion 2005-04 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Ocular comfort/tolerability | Day 1, 3, 8, 15, 22 and 29
Intraocular pressure measurements | Day 1, 3, 8,15, 22 and 29

SECONDARY OUTCOMES:
Assessment of safety | Througout 28-day study

CONTACTS AND LOCATIONS:
Overall Officials: Timothy L Comstock, DO, Study Director — Bausch & Lomb Incorporated

REFERENCES:
- [Derived] Bartlett JD, Holland EJ, Usner DW, Paterno MR, Comstock TL. Tolerability of loteprednol/tobramycin versus dexamethasone/tobramycin in healthy volunteers: results of a 4-week, randomized, double-masked, parallel-group study. Curr Med Res Opin. 2008 Aug;24(8):2219-27. doi: 10.1185/03007990802231981. Epub 2008 Jun 23. PMID 18577309